CLINICAL TRIAL: NCT02010372
Title: Optimizing the Practical Application of Immunization Information System Use in Primary Care Practices
Brief Title: Optimizing Application And Support Of Immunization Information Systems (OASIS)
Acronym: OASIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Stanley J Schaffer, MD, Principal Investigator, University of Rochester
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: 5U01IP000502 (NIH)
Record Dates: First submitted 2013-12-09; First posted 2013-12-12 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2016-02

CONDITIONS: Increase in Use of Immunization Registry; Increase in HPV Vaccination Rate
Keywords: Immunization Registry; Human Papillomavirus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Reminder Recall Reports (Experimental): Training in how to use reminder-recall reports in the Immunization registry will be given to administrators who will then be asked to regularly run these reports for a period of one year.
  Interventions: Other: Reminder Recall Report
- Audit-Feedback/Immunization Forecasting Reports (Experimental): Training in how to use audit-feedback/immunization forecasting reports in the Immunization registry will be given to administrators who will then be asked to regularly run these reports for a period of one year.
  Interventions: Other: Audit-Feedback/Immunization Forecasting Reports
- Control (No Intervention): No intervention will be administered to this group.

INTERVENTIONS:
Other: Reminder Recall Report — Practices (administrators) that are randomized to this intervention will receive training in how to run reminder recall reports for patients due to receive any dose of HPV vaccine. After the training has been completed, administrators will be asked to continue running regularly scheduled reports over the course of one year. A tracking log will be sent regularly to the research team.
  Arms: Reminder Recall Reports
Other: Audit-Feedback/Immunization Forecasting Reports — Practices (administrators) that are randomized to this intervention will receive training in how to run audit-feedback/immunization forecasting reports for patients due to receive any dose of HPV vaccine and to determine the % of patients in their practice who have received at least one dose of HPV vaccine within the study period. After the training has been completed, administrators will be asked to continue running regularly scheduled reports over the course of one year. A tracking log will be sent regularly to the research team.
  Arms: Audit-Feedback/Immunization Forecasting Reports

SUMMARY:
The overall purpose of this study is to evaluate the use of features of the New York State Immunization Information System (NYSIIS) by various types of primary care practices and determine how best to promote the use of IIS features and functionality. The primary goal is to promote the use of NYSIIS for immunization quality improvement (QI) in the practice setting. Customized training sessions will be conducted by study staff to educate practices on NYSIIS' enhanced features.

ELIGIBILITY:
Inclusion Criteria:

* NYSIIS administrator at a participating practice

Exclusion Criteria:

* Practices already utilizing/running reports used in the intervention

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2013-12; Primary Completion 2015-05 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
NYSIIS report usage | One Year
  Practice NYSIIS administrators will monitor the number of reports their practice generates throughout the 12 month post-training period. These measures for control and intervention practices will be compared in bivariate and multivariate analysis.

SECONDARY OUTCOMES:
HPV Vaccination Rate | One Year
  HPV Vaccination rates will be measured to determine the change in the practice's immunization levels (for the pre-determined immunization QI goal) over the 12-month period following their initial training. Statistical comparisons of control and intervention practice will be performed using bivariate analyses, while multivariate analyses will be used to account for the effects of practice characteristics.

CONTACTS AND LOCATIONS:
Overall Officials: Stanley J Schaffer, MD, MPH, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States